CLINICAL TRIAL: NCT00298493
Title: A Randomized Trial of Daily Sedative Interruption in Critically Ill Patients Being Managed With a Sedation Protocol - A Pilot Study
Brief Title: Daily Sedative Interruption in Critically Ill Patients Being Managed With a Sedation Protocol
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MSH REB#00-0032-A
Record Dates: First submitted 2006-02-28; First posted 2006-03-02 (Estimated); Last update posted 2006-03-02 (Estimated); Status verified 2006-02

CONDITIONS: Critical Illness; Mechanical Ventilation
Keywords: ICU; Sedation strategies; Daily sedative interruption; Sedation protocols
MeSH Terms: conditions — Critical Illness

INTERVENTIONS:
Procedure: Sedation management strategy

SUMMARY:
All critically ill, mechanically ventilated patients in the Intensive Care Unit receive medications to relieve pain and anxiety. However, accumulation of these medications can be associated with serious complications, most notably longer time on the breathing machine and in the ICU. Two strategies have been shown to dramatically improve patient outcomes: nurse-directed protocols for giving sedation, and daily interruption of sedation. However, these strategies have not been widely adopted, because of physicians' concerns, and because it is unclear which strategy is better. Given that patient outcome is improved with either of these strategies, the fundamental question that arises is whether patients managed with a combination of two strategies which both reduce drug accumulation (protocolized sedation and daily interruption) have an even better outcome than patients managed with only one of them (protocolized sedation). We propose a multicenter study in which 700 critically ill, mechanically ventilated patients will have their sedation managed with protocolized sedation alone, or both strategies. Both groups of patients will have the following recorded: ICU and hospital lengths of stay, mortality, total sedative drug use, ICU human resources used, side effects and recall of their ICU stay. The results of this large multi-center trial will help to inform best practice with regard to sedation management of critically ill patients in Canada and elsewhere. In addition, reducing ICU stay could be economically attractive, as the cost of an ICU day in Canada is approximately $3000.

ELIGIBILITY:
Inclusion Criteria:

1. age>18 years
2. Mechanically ventilated, with anticipated need for MV ≥ 48 hours
3. ICU team has decided to initiate continuous sedative/analgesic infusion(s)
4. informed consent.

Exclusion Criteria:

1. Admission after resuscitation from cardiac arrest
2. Traumatic brain injury
3. Currently receiving neuromuscular blocking agents
4. Allergy to any of the study medications
5. History of alcohol, sedative or analgesic abuse
6. History of psychiatric illness
7. Acute or chronic neurologic dysfunction
8. Administration of sedatives for >24 hr,
9. Lack of commitment to aggressive treatment
10. Current enrollment in a related trial
11. Previous enrollment in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65
Dates: Start 2001-02; Study Completion 2004-09

PRIMARY OUTCOMES:
Duration of Mechanical Ventilation
ICU and Hospital Lengths of stay

SECONDARY OUTCOMES:
Adverse events
Patient Recall
Caregiver workload

CONTACTS AND LOCATIONS:
Overall Officials: Sangeeta Mehta, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Mehta S, Burry L, Martinez-Motta JC, Stewart TE, Hallett D, McDonald E, Clarke F, Macdonald R, Granton J, Matte A, Wong C, Suri A, Cook DJ; Canadian Critical Care Trials Group. A randomized trial of daily awakening in critically ill patients managed with a sedation protocol: a pilot trial. Crit Care Med. 2008 Jul;36(7):2092-9. doi: 10.1097/CCM.0b013e31817bff85. PMID 18552687